CLINICAL TRIAL: NCT03175146
Title: Stereotactic Body RadioTherapy (SBRT) for Oligo-metastatic Colo-rectal Cancer With Bio-marker Evaluation for Early Progression
Brief Title: A Study to See Whether Stereotactic Body RadioTherapy (SBRT) Can Shrink Tumours Within the Liver Safely
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC L-SBRT 15-01
Record Dates: First submitted 2016-01-06; First posted 2017-06-05 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Colonic Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Stereotactic Body Radiation Therapy
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — 5 treatments given over 2 weeks
  Other Names: SBRT

SUMMARY:
The proposed study will evaluate if "curative intent" SBRT can provide high response rates and clinically meaningful cancer control with acceptable toxicity specifically in patient with metastatic colorectal cancer (mCRC) who do not have surgical options and are no longer responding to systemic therapy

DETAILED DESCRIPTION:
SBRT for Oligo-metastatic Colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Colo-rectal Cancer
* 1-3 Liver metastasis measurable on Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
* Surgically resected primary disease
* Technically/medically inoperable or patient declined surgery
* Progression or Stability after at least 1 Line of chemotherapy
* Adequate marrow function: Hb > 80g/L, Platelets > 100 x 109/L, White blood cell > 2 x 109/L
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Age > 18 years
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

* Prior liver radiation, or radiation in close proximity to planned treatment sites
* Prior invasive malignancy
* Severe, active co-morbidity
* Active hepatitis or Child Pugh Score B (9) or worse
* Pregnant or nursing women
* Extra hepatic disease: Any Bone/Any Brain, 2 or more Lung metastasis
* Life expectancy < 6 mo from any cause
* Concurrent chemotherapy
* Response to prior chemotherapy with minimal measurable disease in liver

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Response rate within the treated liver lesion | 6 months
  RECIST Response

SECONDARY OUTCOMES:
Progression-free survival | Up to 5 years
  Any progression of the disease
Toxicity | From date of randomization up to 5 years
  Grade 3 CTCAE events
Quality of Life | From date of Randomization to Death or Progression or 5 years whichever comes first.
  Fact - H quality of life instrument
Median survival | From date of randomization upto 5 years
  Median survival
Overall survival | From date of randomization upto 5 years
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Richie Sinha, MD, Principal Investigator — Tom Baker Cancer Centre

IPD SHARING:
Plan to Share IPD: Yes